CLINICAL TRIAL: NCT01148550
Title: Longitudinal Study of Mitochondrial Hepatopathies
Acronym: MITOHEP
Status: Suspended | Type: Observational
Sponsor: Arbor Research Collaborative for Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: MITOHEP Study-ChiLDReN Network; U01DK103149 (NIH); U01DK103140 (NIH); U01DK103135 (NIH); U01DK084575 (NIH); U01DK084538 (NIH); U01DK084536 (NIH); U01DK062503 (NIH); U01DK062500 (NIH); U01DK062497 (NIH); U01DK062481 (NIH); U01DK062470 (NIH); U01DK062466 (NIH); U01DK062456 (NIH); U01DK062453 (NIH); U01DK062452 (NIH); U01DK062445 (NIH); U01DK062436 (NIH); U24DK062456 (NIH)
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Last update posted 2025-10-15 (Actual); Status verified 2025-08

CONDITIONS: Acute Liver Failure; Mitochondrial Diseases; End Stage Liver Disease; Respiratory Chain Deficiencies, Mitochondrial; Disorder of Fatty Acid Oxidation
Keywords: neonatal acute liver failure; late-onset liver failure; cholestasis,; fatty liver,; liver dysfunction,; cirrhosis
MeSH Terms: conditions — Liver Failure, Acute; Mitochondrial Diseases; End Stage Liver Disease; Cholestasis; Fatty Liver; Liver Diseases; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group 1: Mitochondrial Hepatopathy Disease Group

SUMMARY:
The specific aims of this study are (1) to determine the clinical phenotypes and natural history of hepatic RC and FAO disorders, (2) to determine the correlation between genotype and phenotype, (3) to determine if circulating biomarkers reflect diagnosis and predict liver disease progression and survival with the native liver, (4) to determine the clinical outcome of these disorders following liver transplantation, and (5) to develop a repository of serum, plasma, urine, tissue and DNA specimens that will be used in ancillary studies. To accomplish these aims, the ChiLDReN investigators at clinical sites (currently 9 sites) will prospectively collect defined data and specimens in a uniform fashion at fixed intervals in a relatively large number of subjects. Clinical information collected from subjects and their parents will enhance the potential for meaningful research in these disorders. A biobank of previously collected subject specimens and DNA samples will be established for use in ancillary studies to be performed in addition to this study.

DETAILED DESCRIPTION:
This study will be conducted as part of the NIH-supported Childhood Liver Disease Research and Education Network (ChiLDREN). ChiLDREN is investigating rare cholestatic liver diseases of childhood: alpha-1 antitrypsin deficiency (A1AT), Alagille's Syndrome (AGS), progressive familial intrahepatic cholestasis (PFIC), bile acid synthesis defects and mitochondrial hepatopathies (all previously studied by the Cholestatic Liver Disease Consortium [CLiC]); biliary atresia (previously studied by the Biliary Atresia Research Consortium [BARC]); neonatal hepatitis; and cystic fibrosis liver disease, which is studied by a new branch of ChiLDREN known as the Cystic Fibrosis Liver Disease (CFLD) Network.

In this protocol, mitochondrial hepatopathies in children and young adults will be investigated. The focus will be on respiratory chain defects (RC) and defects of fatty acid oxidation (FAO). There is little known about the full spectrum of severity and long-term natural history of mitochondrial hepatopathies. Moreover, these disorders have not been subject to prospective, rigorous clinicopathological scrutiny.

ELIGIBILITY:
Subjects in Group 1 (Mitochondrial Hepatopathy group) must meet all of the following inclusion criteria:

1. Children and young adults with suspected or documented hepatic RC defector FAO defect from birth to 18 years old (through 18 years).
2. Both sexes, all races and ethnic groups.
3. Participants must meet one of the following sets of criteria (A or B):

A. Potential subjects presenting with acute or chronic liver disease or acute liver failure but who have not had a liver transplant must meet one of Clinical Criteria 1 and one of Clinical Criteria 2 listed below:

1. Clinical Criteria 1 (any one of the following)

   * 1.Acute liver failure, defined as severe liver dysfunction and either 1) INR >1.5 or prothrombin time > 15 seconds with encephalopathy or 2) INR > 2.0 or prothrombin time > 20 seconds with or without encephalopathy; occurring within 8 weeks of onset of illness; with no known underlying chronic liver disease, or
   * 2.Acute liver disease defined as elevated AST or ALT >1.25 ULN and CK <1000u/L or conjugated bilirubin >2.0 mg/dl and >20% of total bilirubin, or
   * 3.Chronic liver disease defined as:

     * elevated ALT or AST (>1.25 ULN) for > 6 months, or
     * conjugated hyperbilirubinemia (conjugated [direct] > 2.0 mg/dl and > 20% of total bilirubin) for > 6 months or
     * clinical stigmata of chronic liver disease, including chronic hepatomegaly, clinical findings or complications of cirrhosis or portal hypertension, impaired liver synthetic function, intractable pruritus explainable only by liver disease or end-stage liver disease, or
     * abnormal liver histology including hepatic fibrosis or cirrhosis, microvesicular steatosis, canalicular cholestasis, ballooned granular red hepatocytes (AKA oncocytes), intralobular collapse/regeneration And
2. Clinical Criteria 2 (any one of the following):

   * 1.Prior history of extra-hepatic organ involvement accompanied by any one or more of the signs and symptoms associated with mitochondrial dysfunction (e.g.

hypotonia, neuro-developmental delay, seizure disorder requiring treatment with valproic acid, nystagmus, cardiomyopathy, renal tubulopathy, bone marrow failure, myopathy, hearing loss), or

* 2.Lactic acidosis (arterial blood or free-flowing venous blood level >2.5 mmol/L or >22.5 mg/dl at any age and increased lactate:pyruvate ratio [>25.0]) or
* 3.Hypoglycemia (blood glucose <45 mg/dl on any measurement) and hypoketonuria (<1+ for urine ketones by dipstick on urine specimen obtained within 4 hours after collecting blood with low glucose concentration), or
* 4.Abnormal acyl carnitine profile, or
* 5.Documented biochemical (enzymatic) or genetic diagnosis

B. Potential participants who have undergone a liver transplantation because of acute liver failure or end stage liver disease due to suspected or confirmed mitochondrial hepatopathy; the transplantation may have been performed at a non-ChiLDREN medical center or at a ChiLDREN Clinical Site. Participants will meet Criteria 1 and either criteria 2 or criteria 3 below:

* 1.Previous liver transplantation, AND
* 2.Suspected mitochondrial liver disease, based upon meeting one or more of the following criteria:

  * Had a prior history of extra-hepatic organ involvement accompanied by signs and symptoms associated with mitochondrial dysfunction (e.g., hypotonia, neuro-developmental delay, seizure disorder requiring treatment with valproic acid, nystagmus, cardiomyopathy, renal tubulopathy, bone marrow failure, myopathy, hearing loss), OR
  * A prior history of lactic acidosis (arterial blood or free-flowing venous blood level >2.5 mmol/L or >22.5 mg/dl at any age and increased lactate:pyruvate ratio [>25.0]), OR
  * A prior history of hypoglycemia (blood glucose <45 mg/dl on any measurement) and hypoketonuria (≤1+ for urine ketones by dipstick on urine specimen obtained within 4 hours after collecting blood with low glucose concentration), OR
  * A prior history of an abnormal acyl carnitine profile, OR
  * Documented biochemical (enzymatic) or genetic diagnosis of a mitochondrial disorder
* 3.A documented (confirmed) mitochondrial disorder based upon the confirmation criteria specified in protocol.

Subjects in Group 2 (Suspected Mitochondrial Hepatopathy not meeting Group 1 enrollment criteria) must meet the following inclusion criteria:

1. Children and young adults with suspected hepatic RC defect or FAO defect between birth through 18 years but who do not meet clinical inclusion criteria listed above for acute or chronic liver disease or acute liver failure.
2. Both sexes, all races and ethnic groups.

Subjects in either Group 1 or 2 must not have any of the following exclusion criteria:

1. Inability to comply with the longitudinal follow-up described below.
2. Failure of a family/patient to sign the informed consent/assent document or the HIPAA authorization form.
3. Known Medium Chain Acyl CoA Dehydrogenase deficiency (MCAD).
4. Other known causes of liver disease.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of 150 children and young adults with suspected or documented hepatic RC defect or FAO defect between birth and 18 years old from both genders and all races and ethnic groups that meet inclusion/exclusion criteria as defined above
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2010-08-18 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Listing for liver transplant | Measured/assessed at baseline, 6 months, Years 1 through 10, and at time of liver transplant, liver or muscle biopsy or hospitalization for critical illness if applicable
  Listing for liver transplant
Liver transplantation | Measured/assessed at baseline, 6 months, Years 1 through 10, and at time of liver transplant, liver or muscle biopsy or hospitalization for critical illness if applicable
  Liver transplantation
Involvement of other organ systems known to be associated with mitochondrial diseases | Measured/assessed at baseline, 6 months, Years 1 through 10, and at time of liver transplant, liver or muscle biopsy or hospitalization for critical illness if applicable
  Involvement of other organ systems known to be associated with mitochondrial diseases
Death | Measured/assessed at baseline, 6 months, Years 1 through 10, and at time of liver transplant, liver or muscle biopsy or hospitalization for critical illness if applicable
  Death

SECONDARY OUTCOMES:
Growth failure | Measured/assessed at baseline, 6 months, Years 1 through 10, and at time of liver transplant, liver or muscle biopsy or hospitalization for critical illness if applicable
  Growth failure (defined as weight or length Z-score for age < -2)
Worsening liver function | Measured/assessed at baseline, 6 months, Years 1 through 10, and at time of liver transplant, liver or muscle biopsy or hospitalization for critical illness if applicable
  Worsening liver function (defined as PELD >10)
Complications of portal hypertension | Measured/assessed at baseline, 6 months, Years 1 through 10, and at time of liver transplant, liver or muscle biopsy or hospitalization for critical illness if applicable
  Complications of portal hypertension
Neurodevelopmental outcome | Measured/assessed at baseline, 6 months, Years 1 through 10, and at time of liver transplant, liver or muscle biopsy or hospitalization for critical illness if applicable
  Neurodevelopmental outcome
Health related Quality of Life | Measured/assessed at baseline, 6 months, Years 1 through 10, and at time of liver transplant, liver or muscle biopsy or hospitalization for critical illness if applicable
  Health related Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Sokol, MD, Study Chair — University of Colorado, Denver; Ed Doo, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); John C Magee, MD, Principal Investigator — University of Michigan; Lisa Henn, PhD, Principal Investigator — Arbor Research Collaborative for Health - Data Coordinating Center; Katrina Loh, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (16):
- United States (15):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California at San Francisco (UCSF), San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta - Emory University, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital (Baylor College of Medicine), Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The data will be transferred to NIDDK at the end of the study.

REFERENCES:
- See also: Childhood Liver Disease Research Network (ChiLDReN) website — https://childrennetwork.org/